CLINICAL TRIAL: NCT03096912
Title: A Phase II Single Arm Study Assessing Efficacy & Safety of Ribociclib in Patients With Advanced Well-Differentiated or Dedifferentiated Liposarcoma
Brief Title: A Study Assessing Efficacy & Safety of Ribociclib in Patients With Advanced Well/Dedifferentiated Liposarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Daniela Katz M.D, M.D, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243/16
Record Dates: First submitted 2016-11-29; First posted 2017-03-30 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Liposarcomas, Dedifferentiated; Liposarcoma - Well Differentiated; Liposarcoma; Mixed Type; Soft-Tissue Sarcoma
Keywords: CDK4 inhibitor; LEE011; ribociclib; liposarcoma dedifferentiated; liposarcoma well differentiated
MeSH Terms: conditions — Liposarcoma; Lipoma; Liposarcoma, Myxoid; Sarcoma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ribociclib (Experimental): Oral, ribociclib 600 mg x 1 a day, 21 days on 7 days off
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — Ribociclib Oral 600 mg x 1 a day 21 days on 1 week off in 28 days cycles
  Other Names: LEE011

SUMMARY:
The purpose of this study is to determine whether ribociclib are effective and safe in the treatment of progressive well/dedifferentiated liposarcoma (WDL/DDL).

DETAILED DESCRIPTION:
The expected duration of this study is 36 months (24 months accrual period and 12 month follow up period). Enrollment into the screening or treatment phase of the study will be stopped when the actual subject numbers have been achieved.

This single arm single institution, open label, prospective, phase II trial will evaluate the efficacy and safety of oral 600mg/daily in 28 day cycles of ribociclib in advanced well-differentiated liposarcoma (WDL) and de-differentiated liposarcoma (DDL) patients. Number of patients in the study will reflect the reconciliation between statistical requirements and incidence.

Treatment will continue until disease progression, development of unacceptable toxicity, noncompliance or withdrawal of consent by the patient or investigator decision.

All screening requirements must be completed within 28 days of the visit (except for CDK4/6 amplification and pRb, p16 and cyclin D staining status which may be completed in advance). Patients will be examined on cycle 1 day-1 and every 2 weeks, including complete blood count (CBC) and chemistry, for the first 8 weeks of treatment, and thereafter every month until disease progression. CT/MRI imaging (contrast) will be performed every 8 weeks for response evaluation. Clinical benefit as well as individual categories of response (complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) will be determined using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST). Response duration endpoints, including PFS, PFS at 12 weeks and OS will be assessed using the Kaplan-Meier method. Toxicity (AEs) will be recorded using the NCI- Common Toxicity Criteria for Adverse Effects v 4.03 (NCI-CTCAE). Screening procedures will include medical history, physical examination, blood test, baseline CT/MRI imaging and formalin-fixed tissue submission for FoundationOne mutational analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Histological confirmed diagnosis of WDL/DDL with metastatic or locally advanced disease not amenable to complete resection
* WDL/DDL patients must have documentation of disease progression within 6 months prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Measurable disease by RECIST v1.1 criteria. At least one measurable lesion located outside of a previously irradiated area
* Formalin fixed paraffin embedded tumor blocs and representative hematoxylin/eosin slides (preferably both) should be provided for immunohistochemistry staining and molecular analysis of 50 gene signature panel and must have increased CDK4 gene copy number (at least >/=3) and proficient Rb gene
* Patient has adequate bone marrow and organ function
* Must be able to swallow ribociclib capsules/tablets

Exclusion Criteria:

* A known hypersensitivity to ribociclib or any of its excipients
* A concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer
* Patients with central nervous system (CNS) involvement at least 4 weeks from prior therapy completion
* Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening)
* On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 msec
* Participation in a prior investigational study within 30 days prior to enrollment
* Patient has had major surgery within 14 days prior to starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Response to therapy as evaluated by RECIST 1.1 | 36 months
Response to therapy as evaluated by Choi | 36 months

SECONDARY OUTCOMES:
Median PFS | 36 months
  PFS will be computed from the date of start of treatment to the first documented date of progression or the date of death, due to any cause assessed by investigator.
PFS assessed at 12 weeks | 12 weeks
  Number of total patients who are PFS at 12 weeks of treatment
Overall survival (OS) | 36 months
  will be computed from the date of start of treatment to the date of death, due to any cause. Patients alive or lost for follow-up at the time of the analysis will be censored at the date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Katz, M.D, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No